CLINICAL TRIAL: NCT05932069
Title: The Active AMD Study to Improve Function in Veterans With Age Related Macular Degeneration
Brief Title: Active AMD Study to Improve Function in Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C4563-R; 1I01RX004563 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-07-06 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Age Related Macular Degeneration (AMD)
Keywords: Age Related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPIN (Experimental): Exercise 3 times a week on a stationary ergometer @ 50-80% of maximal heart rate reserve for 20 minutes to 45 minutes per session
  Interventions: Behavioral: SPIN
- Non-aerobic, stretching/balance intervention Control (Active Comparator): For this arm of the intervention, randomized participants followed the same guidelines as the SPIN group but did not partake in aerobic exercise. To equalize contact/monitoring of the groups this group met for the same total duration time as the SPIN group; however, instead of aerobic exercise, progressive whole body stretching and toning exercises
  Interventions: Behavioral: Non-aerobic, stretching/balance intervention Control

INTERVENTIONS:
Behavioral: SPIN — Stationary cycling
  Arms: SPIN
Behavioral: Non-aerobic, stretching/balance intervention Control — Balance and stretching exercise
  Arms: Non-aerobic, stretching/balance intervention Control

SUMMARY:
Age Related Macular Degeneration (AMD) is the leading cause of vision loss among Veterans aged 50 years and older. AMD also adversely affects mortality, physical and cognitive functioning, and activities of daily living. These debilitations negatively impact quality of life for US Veterans. Unfortunately, there are no cures and few treatments. With the increase in the aging Veteran population and the increasing prevalence of AMD, it is imperative to identify and implement strategies to limit the functional burden of AMD. To address this growing challenge, the investigators propose to test the impact of a proven exercise intervention, stationary bicycling (spinning), on visual and non-visual negative health outcomes in AMD. The work in several retinal degeneration mouse models shows that aerobic exercise significantly preserves retinal morphology and function and visual acuity. Even more exciting, the investigators' preliminary work with older Veterans with and without AMD suggests that spin cycling modestly but significantly benefits visual acuity in aged Veterans. Based on this work, the investigators propose to implement a 6-month synchronous, online group spin cycling program for Veterans with AMD, evaluating effects on physical, cognitive, and visual outcomes.

DETAILED DESCRIPTION:
Aim 1 is to determine if exercise training preserves visual outcomes in Veterans with intermediate AMD when compared to a non-aerobic exercised, contact-controlled AMD group. Best corrected visual acuity, dark adaptometry, contrast sensitivity, optical coherence tomography angiography (OCT-A) and the Low Luminance Questionnaire will be assessed before, mid, and after the 6-month interventional period. In line with previous animal and human subject studies, the investigators also hypothesize a correlation between improved visual function with increases in serum brain derived neurotrophic factor (BDNF). Aim 2 is to determine if exercise improves physical and cognitive function in Veterans with AMD when compared to non-aerobic exercised, contact-controlled AMD group. The investigators will test the timed-up-and-go (TUG) and a neuropsychological battery, mid- and post 6-month interventional period. These provide a robust index of other health, well-being, and quality of life related outcomes in numerous older adult patient populations. In line with the preliminary studies, the investigators' working hypothesis is that 6 months of exercise will result in a clinically significant improvement in TUG performance as well as improved cognitive-executive functions. The investigators expect that the results from achieving these aims will set the stage for a larger, multi-site trial powered to test the hypothesis that virtual exercise can slow the progression of AMD while improving physical and cognitive function and quality of life in Veterans. Thus, the investigators propose an accessible, low-cost intervention that can be easily scalable to other VA centers to improve engagement/adherence, while also improving visual and functional capacity for Veterans with AMD who are at high risk for comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit Veterans with a diagnosis of intermediate stage AMD in at least one eye, aged 65-89, willing and able to cooperate with assessments and interventions.
* Eligible participants will be quantified > 26 on the Montreal Cognitive Assessment (MoCA) to meet the criteria for cognitively intact.
* Participants will be free from diseases affecting cognition or ability to engage in aerobic exercise (including but not limited to chronic heart, liver, or kidney disease) and from diseases/injuries directly affecting brain functions (including but not limited to significant closed head injury, open intracranial wounds, stroke, epilepsy, degenerative diseases of the nervous system).
* Eligible participants will be required to have stable internet access in their home.
* All subjects will speak English as a primary language and will have graduated high school so that behavioral/cognitive measures reflect effects of age, AMD, and/or aerobic exercise and not the effects of familiarity with English or lack of education.

Exclusion Criteria:

* Other, non-AMD, visual impairments. Potential participants with major psychiatric disorder (including but not limited to psychosis, major depression, bipolar disorder) by history will be excluded as well as individuals with current alcohol or substance use disorder.
* Additionally, individuals with cardiovascular disease and or history of myocardial infarction will not be included.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
contrast sensitivity | Change from Baseline contrast sensitivity at 6 months
  1.Contrast Sensitivity (CS) will be determined using the CSV1000E Contrast Chart. This test provides for four rows ofsine-wave gratings. Subjects will view the chart from a distance of 2.5m. Subjects will view the chart monocularly while wearing their normal correction. CS thresholds will be assessed for both eyes individually.
Dark adaptometry | Change from Baseline dark adaptometry at 6 months
  Dark adaptometry (primary vision outcome measure). Dark adaptation or night vision is known to be affected with increasing stages of AMD. This test probes the ability of the eye to dark adapt. Participants will be asked to place their head on a chin rest in front of the machine. Each eye will be tested individually, and the opposing eye will be covered with an eye patch. While fixating on a light at the back of the machine, a bright flash will be presented to bleach the photoreceptors and then a series of dimmer flashes will appear and the participant will be asked to identify whether or not they saw the flashes by pushing a response button. The duration of the test is ~7 minutes per eye.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | Change from best corrected visual acuity at 6 months
  Best Corrected Visual Acuity (BCVA) is measured using the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart Subjects will be placed at a distance of 4 m, if at least the top line can be read correctly, and encouraged to give a response for each letter until 5 successive incorrect answers are recorded. This test will take 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Joe R. Nocera, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bello MO, Mammino KM, Vernon MA, Wakeman DG, Denmon CA, Krishnamurthy LC, Krishnamurthy V, McGregor KM, Novak TS, Nocera JR. Graded Intensity Aerobic Exercise to Improve Cerebrovascular Function and Performance in Older Veterans: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 26;13:e58316. doi: 10.2196/58316. PMID 39326042